CLINICAL TRIAL: NCT00239577
Title: Observer-blind, Single Center, Controlled Study of 2 Doses of Various Formulations of the WRAIR Live Attenuated Tetravalent Dengue Vaccine Compared to a Placebo Control, Administered on a 0-6-month Schedule, to Healthy Adults
Brief Title: A Trial of a Walter Reed Army Institute of Research (WRAIR) Live Attenuated Virus Tetravalent Dengue Vaccine in Healthy US Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 103996
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Dengue
Keywords: Dengue infection
MeSH Terms: conditions — Dengue

ARMS (4):
- DENGUE FORMULATION 17A GROUP (Experimental): Healthy male or female subjects, between and including 18-45 years of age, who received two doses of Dengue vaccine Formulation 17a, administered subcutaneously into the upper-outer triceps/deltoid area of the non-dominant arm, at Months 0 and 6.
  Interventions: Biological: Live attenuated tetravalent dengue vaccine
- DENGUE FORMULATION 17B GROUP (Experimental): Healthy male or female subjects, between and including 18-45 years of age, who received two primary doses of Dengue vaccine Formulation 17b, administered subcutaneously into the upper-outer triceps/deltoid area of the non-dominant arm, at Months 0 and 6, and one booster dose approximately 5-12 months after the second dose.
  Interventions: Biological: Live attenuated tetravalent dengue vaccine
- DENGUE FORMULATION 19 GROUP (Experimental): Healthy male or female subjects, between and including 18-45 years of age, who received two primary doses of Dengue vaccine Formulation 19, administered subcutaneously into the upper-outer triceps/deltoid area of the non-dominant arm, at Months 0 and 6 and one booster dose approximately 5-12 months after the second dose.
  Interventions: Biological: Live attenuated tetravalent dengue vaccine
- PLACEBO GROUP (Placebo Comparator): Healthy male or female subjects, between and including 18-45 years of age, who received two doses of Placebo, administered subcutaneously into the upper-outer triceps/deltoid area of the non-dominant arm, at Months 0 and 6.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Live attenuated tetravalent dengue vaccine — Live attenuated tetravalent dengue vaccine
  Arms: DENGUE FORMULATION 17A GROUP; DENGUE FORMULATION 17B GROUP; DENGUE FORMULATION 19 GROUP
Biological: Placebo — Placebo
  Arms: PLACEBO GROUP

SUMMARY:
This descriptive study will evaluate the safety and immunogenicity of 5 different formulations of the WRAIR dengue vaccine compared to a placebo.

DETAILED DESCRIPTION:
Subjects will be randomized into one of 6 groups. One group will receive a placebo vaccine and the others will receive one of 5 different dengue vaccine formations. Each subject will receive two doses six months apart. Study subjects who elect to participate in a mosquito transmissibility component of the study will undergo mosquito feedings during each of the two assigned follow-up visits after vaccine dose 1. All subjects will have 11 venipunctures during 11 visits (i.e., screening plus 10 study visits) over a period of nine months.

ELIGIBILITY:
Inclusion:

* Healthy male or female adult 18-45 years at the time of vaccination
* Free of obvious health problems as established by medical history and physical examination before entering into the study
* Written informed consent obtained from the subject
* Able to read the Subject Information Sheet and Consent Form
* Subjects who the investigator believes can and will comply with the requirements of the protocol
* Females must be of non-childbearing potential, or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions as defined in the protocol for 30 days prior to vaccination, have a negative pregnancy test within 48 hours prior to vaccination and must agree to continue such precautions for 60 days after completion of the vaccination series

Exclusion:

History of:

* recurrent migraine headache
* any neurological or behavioral disorder or seizures
* drug abuse or alcohol consumption (more than 2 drinks per day)
* allergic disease/reaction likely to be exacerbated by vaccine
* urticaria related to mosquito bites requiring medical attention
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, renal, hematologic or endocrine functional defect
* Any confirmed or suspected immunosuppressive or immunodeficient condition;
* Seropositive for HBsAg, anti-HCV or anti-HIV
* Acute disease at the time of enrollment
* Chronic hepatomegaly or splenomegaly
* Use of any investigational or non-registered drug or vaccine within 30 days preceding study or planned use
* Planned administration of a vaccine not foreseen by the study protocol 30 days ±each vaccine dose
* Planned move during study
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs or administration of immunoglobulins and/or blood products, within 90 days preceding the first dose or planned administration during the study period
* Any chronic systemic drug therapy to be continued during the study period

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2006-04-05 (Actual); Primary Completion 2007-06-19 (Actual); Study Completion 2007-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Silver Spring, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Primary Phase
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Started | 22 | 22 | 21 | 21
Completed | 17 | 19 | 18 | 21
Not Completed | 5 | 3 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Other | 5 | 3 | 2 | 0
Period: Booster Phase
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Started | 0 (The subjects belonging to this group did not receive a booster dose of Dengue vaccine.) | 9 | 12 | 0 (The subjects belonging to this group did not receive an additional dose of Placebo.)
Completed | 0 (The subjects belonging to this group did not receive a booster dose of Dengue vaccine.) | 9 | 12 | 0 (The subjects belonging to this group did not receive an additional dose of Placebo.)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group | Total
Number analyzed (Participants) | 22 | 22 | 21 | 21 | 86
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.90 (7.75) | 32.80 (6.93) | 33.0 (8.60) | 35.8 (6.70) | 34.37 (7.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 8 | 10 | 35
  Male | 16 | 11 | 13 | 11 | 51

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: During the 21-day (Days 0-20) follow-up after Dose 1 of the study vaccine
Population: The analysis was performed on the Primary Total Vaccinated Cohort, which included all vaccinated subjects (with at least one vaccine administration documented) for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 22 | 22 | 21 | 21
Participants
  Any Pain | 7 | 2 | 4 | 5
  Grade 3 Pain | 0 | 0 | 0 | 1
  Any Redness | 8 | 3 | 4 | 4
  Grade 3 Redness | 1 | 1 | 0 | 0
  Any Swelling | 6 | 4 | 5 | 2
  Grade 3 Swelling | 0 | 1 | 1 | 1

2. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were abdominal pain, arthralgia, fatigue, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], headache, muscle aches, nausea, pain behind the eyes, photophobia, pruritus, rash and vomiting. Any = occurrence of the symptom regardless of intensity grade or relation to vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 21-day (Days 0-20) follow-up after Dose 1 of the study vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 22 | 22 | 21 | 21
Participants
  Any Abdominal pain | 0 | 3 | 3 | 4
  Grade 3 Abdominal pain | 0 | 0 | 1 | 0
  Related Abdominal pain | 0 | 2 | 2 | 3
  Any Arthralgia | 5 | 2 | 2 | 3
  Grade 3 Arthralgia | 0 | 0 | 0 | 1
  Related Arthralgia | 4 | 2 | 2 | 2
  Any Fatigue | 8 | 5 | 5 | 7
  Grade 3 Fatigue | 0 | 0 | 1 | 1
  Related Fatigue | 5 | 2 | 4 | 6
  Any Fever | 4 | 2 | 2 | 1
  Grade 3 Fever | 0 | 0 | 0 | 1
  Related Fever | 3 | 2 | 2 | 1
  Any Headache | 12 | 8 | 7 | 7
  Grade 3 Headache | 0 | 0 | 0 | 0
  Related Headache | 8 | 5 | 3 | 5
  Any Muscle aches | 5 | 2 | 3 | 4
  Grade 3 Muscle aches | 0 | 0 | 0 | 2
  Related Muscle aches | 3 | 1 | 3 | 3
  Any Nausea | 5 | 3 | 3 | 1
  Grade 3 Nausea | 0 | 0 | 0 | 0
  Related Nausea | 4 | 0 | 2 | 1
  Any Pain behind eyes | 4 | 4 | 5 | 2
  Grade 3 Pain behind eyes | 0 | 0 | 0 | 0
  Related Pain behind eyes | 4 | 3 | 4 | 2
  Any Photophobia | 3 | 1 | 4 | 2
  Grade 3 Photophobia | 0 | 0 | 0 | 1
  Related Photophobia | 3 | 1 | 3 | 2
  Any Pruritus | 8 | 3 | 2 | 4
  Grade 3 Pruritus | 0 | 0 | 0 | 0
  Related Pruritus | 4 | 2 | 2 | 3
  Any Rash | 4 | 3 | 1 | 0
  Grade 3 Rash | 0 | 0 | 0 | 0
  Related Rash | 4 | 3 | 1 | 0
  Any Vomiting | 2 | 1 | 0 | 0
  Grade 3 Vomiting | 0 | 0 | 0 | 0
  Related Vomiting | 1 | 0 | 0 | 0

3. Primary Outcome: Titers for DEN Neutralizing Antibodies Types 1, 2, 3 and 4
Description: Titers for DEN-1, DEN-2, DEN-3 and DEN-4 neutralizing antibodies, expressed as Geometric Mean Titers (GMTs), with cut-off values greater than or equal to (≥) 10 estimated dose giving 50% (ED50) signal reduction when compared to a control without serum.
Time Frame: At 30 days (Month 7) after Dose 2 of the study vaccine
Population: The analysis was performed on the Primary ATP cohort for immunogenicity, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: ED50
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 16 | 18 | 15 | 19
ED50
  DEN-1 | 241 [81 to 719] | 83 [25 to 273] | 204 [69 to 603] | 7 [4 to 14]
  DEN-2 | 691 [407 to 1175] | 223 [76 to 656] | 342 [123 to 954] | 6 [4 to 10]
  DEN-3 | 94 [28 to 321] | 55 [17 to 177] | 96 [30 to 309] | 6 [4 to 10]
  DEN-4 | 350 [85 to 1439] | 91 [27 to 305] | 84 [24 to 294] | 6 [4 to 8]

4. Primary Outcome: Titers for DEN Neutralizing Antibodies Types 1, 2, 3 and 4 Based on Priming Status
Description: Titers for DEN-1, DEN-2, DEN-3 and DEN-4 neutralizing antibodies, expressed as Geometric Mean Titers (GMTs), with cut-off values greater than or equal to (≥) 10 estimated dose giving 50% (ED50) signal reduction when compared to a control without serum. Not primed = Not primed by MN50; Primed = Primed by MN50. Primed subject is a subject with neutralizing antibody titer ≥ 10 ED50 at pre-vaccination for at least one DEN type. Not primed subject is a subject with neutralizing antibody titer <10 ED50 for any DEN type at pre-vaccination.
Time Frame: At 5 to 12 months post-Dose 2 of the study vaccine
Population: The analysis was performed on the Booster ATP cohort for immunogenicity, which included all evaluable subjects who completed the primary vaccination course, who had received the booster dose according to their random assignment and for whom data concerning immunogenicity outcome measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: ED50
Arm/Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group
Number analyzed (Participants) | 6 | 7
ED50
  DEN-1, Not primed | 15 [4 to 57] | 35 [6 to 187]
  DEN-1, Primed: number analyzed (Participants) | 2 | 2
  DEN-1, Primed | 521 [40 to 6785] | 2430 [2430 to 2430]
  DEN-2, Not primed | 33 [5 to 203] | 30 [6 to 158]
  DEN-2, Primed: number analyzed (Participants) | 2 | 2
  DEN-2, Primed | 346 [0 to 97683203] | 673 [10 to 46541]
  DEN-3, Not primed | 7 [3 to 20] | 12 [4 to 38]
  DEN-3, Primed: number analyzed (Participants) | 2 | 2
  DEN-3, Primed | 426 [0 to 785070000000000] | 1413 [1165 to 1715]
  DEN-4, Not primed | 29 [2 to 521] | 23 [3 to 168]
  DEN-4, Primed: number analyzed (Participants) | 2 | 2
  DEN-4, Primed | 123 [0 to 15158843] | 766 [1 to 959438]

5. Primary Outcome: Titers for DEN Neutralizing Antibodies Types 1, 2, 3 and 4 Based on Priming Status
Description: Titers for DEN 1, DEN 2, DEN 3 and DEN 4 neutralizing antibodies, expressed as Geometric Mean Titers (GMTs), with cut-off values greater than or equal to (≥) 10 estimated dose giving 50% (ED50) signal reduction when compared to a control without serum. Not primed = Not primed by MN50; Primed = Primed by MN50. Primed subject is a subject with neutralizing antibody titer ≥ 10 ED50 at pre-vaccination for at least one DEN type. Not primed subject is a subject with neutralizing antibody titer <10 ED50 for any DEN type at pre-vaccination.
Time Frame: At Month 1 post-booster dose of the study vaccine
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ED50
Arm/Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group
Number analyzed (Participants) | 6 | 7
ED50
  DEN-1, Not primed | 39 [7 to 226] | 73 [19 to 281]
  DEN-1, Primed: number analyzed (Participants) | 2 | 2
  DEN-1, Primed | 672 [55 to 8245] | 2430 [2430 to 2430]
  DEN-2, Not primed | 104 [15 to 720] | 194 [56 to 675]
  DEN-2, Primed: number analyzed (Participants) | 2 | 2
  DEN-2, Primed | 909 [3 to 255163] | 795 [734 to 861]
  DEN-3, Not primed | 34 [5 to 226] | 19 [5 to 69]
  DEN-3, Primed: number analyzed (Participants) | 2 | 2
  DEN-3, Primed | 890 [0 to 13080837] | 1502 [645 to 3498]
  DEN-4, Not primed | 46 [4 to 535] | 31 [4 to 231]
  DEN-4, Primed: number analyzed (Participants) | 2 | 2
  DEN-4, Primed | 215 [99 to 463] | 618 [0 to 2096791]

6. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: as for outcome 1
Time Frame: During the 21-day (Days 0-20) follow-up after Dose 2 of the study vaccine
Population: The analysis was performed on the Primary Total Vaccinated Cohort, which included all vaccinated subjects (with at least one vaccine administration documented) with the symptom sheet filled in and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 16 | 19 | 18 | 20
Participants
  Any Pain | 7 | 1 | 1 | 2
  Grade 3 Pain | 0 | 0 | 0 | 0
  Any Redness | 1 | 0 | 2 | 2
  Grade 3 Redness | 0 | 0 | 0 | 0
  Any Swelling | 1 | 0 | 0 | 1
  Grade 3 Swelling | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: as for outcome 2
Time Frame: During the 21-day (Days 0-20) follow-up after Dose 2 of the study vaccine
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 16 | 19 | 18 | 20
Participants
  Any Abdominal pain | 0 | 3 | 1 | 1
  Grade 3 Abdominal pain | 0 | 0 | 0 | 0
  Related Abdominal pain | 0 | 2 | 0 | 1
  Any Arthralgia | 1 | 2 | 2 | 0
  Grade 3 Arthralgia | 0 | 1 | 0 | 0
  Related Arthralgia | 1 | 2 | 1 | 0
  Any Fatigue | 4 | 4 | 3 | 3
  Grade 3 Fatigue | 0 | 1 | 0 | 0
  Related Fatigue | 3 | 2 | 1 | 1
  Any Fever | 1 | 2 | 1 | 4
  Grade 3 Fever | 0 | 0 | 0 | 0
  Related Fever | 1 | 2 | 0 | 2
  Any Headache | 6 | 5 | 3 | 5
  Grade 3 Headache | 0 | 1 | 1 | 0
  Related Headache | 3 | 4 | 1 | 3
  Any Muscle aches | 1 | 4 | 1 | 0
  Grade 3 Muscle aches | 0 | 1 | 0 | 0
  Related Muscle aches | 1 | 2 | 1 | 0
  Any Nausea | 1 | 3 | 0 | 1
  Grade 3 Nausea | 0 | 0 | 0 | 0
  Related Nausea | 1 | 2 | 0 | 1
  Any Pain behind eyes | 1 | 4 | 1 | 1
  Grade 3 Pain behind eyes | 0 | 0 | 0 | 0
  Related Pain behind eyes | 0 | 2 | 0 | 0
  Any Photophobia | 1 | 2 | 0 | 2
  Grade 3 Photophobia | 0 | 0 | 0 | 0
  Related Photophobia | 1 | 1 | 0 | 1
  Any Pruritus | 2 | 0 | 1 | 1
  Grade 3 Pruritus | 0 | 0 | 0 | 0
  Related Pruritus | 2 | 0 | 1 | 1
  Any Rash | 3 | 0 | 2 | 0
  Grade 3 Rash | 0 | 0 | 0 | 0
  Related Rash | 3 | 0 | 2 | 0
  Any Vomiting | 0 | 1 | 0 | 0
  Grade 3 Vomiting | 0 | 0 | 0 | 0
  Related Vomiting | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: as for outcome 1
Time Frame: During the 21-day (Days 0-20) follow-up after each dose of the study vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 22 | 22 | 21 | 21
Participants
  Any Pain | 9 | 3 | 5 | 5
  Grade 3 Pain | 0 | 0 | 0 | 1
  Any Redness | 8 | 3 | 5 | 5
  Grade 3 Redness | 1 | 1 | 0 | 0
  Any Swelling | 7 | 4 | 5 | 3
  Grade 3 Swelling | 0 | 1 | 1 | 1

9. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: as for outcome 2
Time Frame: During the 21-day (Days 0-20) follow-up after each dose of the study vaccine
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 22 | 22 | 21 | 21
Participants
  Any Abdominal pain | 0 | 5 | 4 | 4
  Grade 3 Abdominal pain | 0 | 0 | 1 | 0
  Related Abdominal pain | 0 | 3 | 2 | 3
  Any Arthralgia | 6 | 4 | 3 | 3
  Grade 3 Arthralgia | 0 | 1 | 0 | 1
  Related Arthralgia | 5 | 4 | 3 | 2
  Any Fatigue | 10 | 8 | 6 | 7
  Grade 3 Fatigue | 0 | 1 | 1 | 1
  Related Fatigue | 7 | 3 | 5 | 6
  Any Fever | 5 | 4 | 3 | 5
  Grade 3 Fever | 0 | 0 | 0 | 1
  Related Fever | 4 | 4 | 2 | 3
  Any Headache | 14 | 9 | 10 | 9
  Grade 3 Headache | 0 | 1 | 1 | 0
  Related Headache | 9 | 6 | 4 | 7
  Any Muscle aches | 6 | 5 | 4 | 4
  Grade 3 Muscle aches | 0 | 1 | 0 | 2
  Related Muscle aches | 4 | 3 | 4 | 3
  Any Nausea | 6 | 4 | 3 | 2
  Grade 3 Nausea | 0 | 0 | 0 | 0
  Related Nausea | 5 | 2 | 2 | 2
  Any Pain behind the eyes | 4 | 7 | 5 | 3
  Grade 3 Pain behind the eyes | 0 | 0 | 0 | 0
  Related Pain behind the eyes | 4 | 5 | 4 | 2
  Any Photophobia | 4 | 3 | 4 | 4
  Grade 3 Photophobia | 0 | 0 | 0 | 1
  Related Photophobia | 4 | 2 | 3 | 3
  Any Pruritus | 9 | 3 | 3 | 4
  Grade 3 Pruritus | 0 | 0 | 0 | 0
  Related Pruritus | 6 | 2 | 3 | 3
  Any Rash | 7 | 3 | 3 | 0
  Grade 3 Rash | 0 | 0 | 0 | 0
  Related Rash | 7 | 3 | 3 | 0
  Any Vomiting | 2 | 2 | 0 | 0
  Grade 3 Vomiting | 0 | 0 | 0 | 0
  Related Vomiting | 1 | 0 | 0 | 0

10. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up after any study vaccine dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 22 | 22 | 21 | 21
Participants | 15 | 10 | 15 | 12

11. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the whole primary phase of the study (from Day 0 up to Month 9)
Population: The analysis was performed on the Primary Total Vaccinated Cohort, included all vaccinated subjects (with at least one vaccine administration documented) for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 22 | 22 | 21 | 21
Participants | 0 | 0 | 1 | 1

12. Secondary Outcome: Number of Subjects With Alert Values for Safety Laboratory Determinations
Description: Among assessed haematological and biochemical parameters were: Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), hematocrit (HC), absolute neutrophil count (NEU) and platelet count (Platelet).
Time Frame: During the 31-day (Days 0-30) follow-up after each vaccine dose (Month 1 and Month 7)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 21 | 22 | 21 | 21
Participants
  ALT, Month 1 | 0 | 0 | 0 | 0
  ALT, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  ALT, Month 7 | 0 | 0 | 0 | 0
  AST, Month 1 | 0 | 0 | 0 | 0
  AST, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  AST, Month 7 | 0 | 0 | 0 | 0
  HC, Month 1 | 0 | 0 | 0 | 0
  HC, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  HC, Month 7 | 0 | 0 | 0 | 0
  NEU, Month 1 | 0 | 0 | 0 | 0
  NEU, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  NEU, Month 7 | 0 | 0 | 0 | 0
  Platelet, Month 1 | 0 | 0 | 0 | 0
  Platelet, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  Platelet, Month 7 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Subjects With Abnormal Findings at Dengue Physical Examination
Description: The abnormal findings at Dengue physical examination included: Rash, Generalized Rash, Skin Hemorrhage, Conjunctival Hemorrhage, Conjunctival Injection, Mucosal Hemorrhage, Lymphadenopathy, Generalized Lymphadenopathy, Hepatomegaly and Splenomegaly. Rash involved < 50% of the body surface; Generalized rash involved at least 50% of the body surface. Generalized lymphadenopathy was defined as palpable lymph nodes in four or more of the following locations: cervical, axillary, inguinal or other, with right and left sides considered as separate locations.
Time Frame: During the 31-day (Days 0-30) follow-up after each vaccine dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 22 | 22 | 21 | 21
Participants
  Rash, Dose 1 | 1 | 0 | 1 | 0
  Generalized Rash, Dose 1 | 0 | 0 | 1 | 0
  Skin Hemorrhage, Dose 1 | 0 | 0 | 0 | 1
  Conjunctival Hemorrhage, Dose 1 | 0 | 0 | 0 | 0
  Conjunctival Injection, Dose 1 | 2 | 0 | 1 | 1
  Mucosal Hemorrhage, Dose 1 | 2 | 1 | 1 | 1
  Lymphadenopathy, Dose 1 | 3 | 3 | 4 | 3
  Generalized Lymphadenopathy,Dose 1 | 0 | 1 | 0 | 1
  Hepatomegaly, Dose 1 | 2 | 3 | 5 | 2
  Splenomegaly, Dose 1 | 0 | 1 | 1 | 1
  Rash, Dose 2: number analyzed (Participants) | 17 | 19 | 18 | 20
  Rash, Dose 2 | 2 | 1 | 2 | 0
  Generalized Rash, Dose 2: number analyzed (Participants) | 17 | 19 | 18 | 20
  Generalized Rash, Dose 2 | 1 | 0 | 1 | 0
  Skin Hemorrhage, Dose 2: number analyzed (Participants) | 17 | 19 | 18 | 20
  Skin Hemorrhage, Dose 2 | 0 | 0 | 0 | 0
  Conjunctival Hemorrhage, Dose 2: number analyzed (Participants) | 17 | 19 | 18 | 20
  Conjunctival Hemorrhage, Dose 2 | 0 | 0 | 0 | 1
  Conjunctival Injection, Dose 2: number analyzed (Participants) | 17 | 19 | 18 | 20
  Conjunctival Injection, Dose 2 | 1 | 1 | 2 | 0
  Mucosal Hemorrhage, Dose 2: number analyzed (Participants) | 17 | 19 | 18 | 20
  Mucosal Hemorrhage, Dose 2 | 0 | 0 | 0 | 0
  Lymphadenopathy, Dose 2: number analyzed (Participants) | 17 | 19 | 18 | 20
  Lymphadenopathy, Dose 2 | 1 | 3 | 5 | 3
  Generalized Lymphadenopathy,Dose 2: number analyzed (Participants) | 17 | 19 | 18 | 20
  Generalized Lymphadenopathy,Dose 2 | 0 | 0 | 0 | 0
  Hepatomegaly, Dose 2: number analyzed (Participants) | 17 | 19 | 18 | 20
  Hepatomegaly, Dose 2 | 1 | 0 | 3 | 3
  Splenomegaly, Dose 2: number analyzed (Participants) | 17 | 19 | 18 | 20
  Splenomegaly, Dose 2 | 0 | 0 | 0 | 2
  Rash, Across | 3 | 1 | 3 | 0
  Generalized Rash, Across | 1 | 0 | 2 | 0
  Skin Hemorrhage, Across | 0 | 0 | 0 | 1
  Conjunctival Hemorrhage, Across | 0 | 0 | 0 | 1
  Conjunctival Injection, Across | 2 | 1 | 2 | 1
  Mucosal Hemorrhage, Across | 2 | 1 | 1 | 1
  Lymphadenopathy, Across | 4 | 6 | 7 | 4
  Generalized Lymphadenopathy,Across | 0 | 1 | 0 | 1
  Hepatomegaly, Across | 2 | 3 | 6 | 4
  Splenomegaly, Across | 0 | 1 | 1 | 2

14. Secondary Outcome: Number of Subjects With Suspected and Confirmed Dengue
Description: The number of subjects with suspected and confirmed Dengue post-vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up after each vaccine dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 22 | 22 | 21 | 21
Participants
  Suspected dengue, Dose 1 | 1 | 0 | 0 | 1
  Confirmed dengue, Dose 1 | 0 | 0 | 0 | 0
  Suspected dengue, Dose 2: number analyzed (Participants) | 17 | 19 | 18 | 20
  Suspected dengue, Dose 2 | 0 | 0 | 0 | 0
  Confirmed dengue, Dose 2: number analyzed (Participants) | 17 | 19 | 18 | 20
  Confirmed dengue, Dose 2 | 0 | 0 | 0 | 0
  Suspected dengue, Across doses | 1 | 0 | 0 | 1
  Confirmed dengue, Across doses | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Subjects With Measurable Dengue Viremia
Description: The number of subjects with measurable dengue viremia at specified timepoints. Negative = Genome equivalent (GEQ)/µL result is equal to zero; Undetermined = GEQ/µL result is below limit of detection (LOD); Positive = GEQ/µL result is ≥ LOD.
Time Frame: During the 31-day (Days 0-30) follow-up after each vaccine dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 22 | 22 | 21 | 21
Participants
  DEN-1 Positive, Dose 1 | 0 | 0 | 0 | 0
  DEN-1 Undetermined, Dose 1 | 2 | 1 | 2 | 1
  DEN-1 Negative, Dose 1 | 18 | 21 | 19 | 20
  DEN-1 Missing, Dose 1 | 2 | 0 | 0 | 0
  DEN-1 Positive, Dose 2 | 0 | 0 | 0 | 0
  DEN-1 Undetermined, Dose 2 | 1 | 2 | 2 | 1
  DEN-1 Negative, Dose 2 | 15 | 17 | 16 | 19
  DEN-1 Missing, Dose 2 | 6 | 3 | 3 | 1
  DEN-1 Positive, Across doses | 0 | 0 | 0 | 0
  DEN-1 Undetermined, Across doses | 3 | 3 | 3 | 2
  DEN-1 Negative, Across doses | 13 | 16 | 15 | 18
  DEN-1 Missing, Across doses | 6 | 3 | 3 | 1
  DEN-2 Positive, Dose 1 | 0 | 0 | 0 | 0
  DEN-2 Undetermined, Dose 1 | 1 | 1 | 0 | 0
  DEN-2 Negative, Dose 1 | 18 | 20 | 19 | 19
  DEN-2 Missing, Dose 1 | 3 | 1 | 2 | 2
  DEN-2 Positive, Dose 2 | 0 | 0 | 0 | 0
  DEN-2 Undetermined, Dose 2 | 0 | 1 | 1 | 0
  DEN-2 Negative, Dose 2 | 15 | 17 | 15 | 18
  DEN-2 Missing, Dose 2 | 7 | 4 | 5 | 3
  DEN-2 Positive, Across doses | 0 | 0 | 0 | 0
  DEN-2 Undetermined, Across doses | 0 | 2 | 1 | 0
  DEN-2 Negative, Across doses | 15 | 16 | 15 | 18
  DEN-2 Missing, Across doses | 7 | 4 | 5 | 3
  DEN-3 Positive, Dose 1 | 0 | 0 | 0 | 0
  DEN-3 Undetermined, Dose 1 | 0 | 0 | 0 | 0
  DEN-3 Negative, Dose 1 | 20 | 22 | 21 | 21
  DEN-3 Missing, Dose 1 | 2 | 0 | 0 | 0
  DEN-3 Positive, Dose 2 | 0 | 0 | 0 | 0
  DEN-3 Undetermined, Dose 2 | 0 | 0 | 0 | 0
  DEN-3 Negative, Dose 2 | 16 | 19 | 18 | 20
  DEN-3 Missing, Dose 2 | 6 | 3 | 3 | 1
  DEN-3 Positive, Across doses | 0 | 0 | 0 | 0
  DEN-3 Undetermined, Across doses | 0 | 0 | 0 | 0
  DEN-3 Negative, Across doses | 16 | 19 | 18 | 20
  DEN-3 Missing, Across doses | 6 | 3 | 3 | 1
  DEN-4 Positive, Dose 1 | 2 | 1 | 0 | 0
  DEN-4 Undetermined, Dose 1 | 1 | 1 | 1 | 0
  DEN-4 Negative, Dose 1 | 17 | 20 | 20 | 21
  DEN-4 Missing, Dose 1 | 2 | 0 | 0 | 0
  DEN-4 Positive, Dose 2 | 3 | 0 | 0 | 0
  DEN-4 Undetermined, Dose 2 | 0 | 0 | 0 | 0
  DEN-4 Negative, Dose 2 | 13 | 19 | 18 | 20
  DEN-4 Missing, Dose 2 | 6 | 3 | 3 | 1
  DEN-4 Positive, Across doses | 5 | 1 | 0 | 0
  DEN-4 Undetermined, Across doses | 1 | 1 | 1 | 0
  DEN-4 Negative, Across doses | 11 | 17 | 17 | 20
  DEN-4 Missing, Across doses | 5 | 3 | 3 | 1

16. Secondary Outcome: Number of Subjects With Safety Laboratory Determinations Outside the Normal Ranges
Description: Among assessed haematological and biochemical parameters were: Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), hematocrit (HC), absolute neutrophil count (NEU) and platelet count (Platelet). Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter.
Time Frame: During the 31-day (Days 0-30) follow-up after each vaccine dose (Month 1 and Month 7)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 21 | 22 | 21 | 21
Participants
  ALT Below, Month 1 | 0 | 0 | 0 | 0
  ALT Above, Month 1 | 1 | 1 | 1 | 2
  ALT Below, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  ALT Below, Month 7 | 0 | 0 | 0 | 0
  ALT Above, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  ALT Above, Month 7 | 0 | 0 | 0 | 0
  AST Below, Month 1 | 0 | 0 | 0 | 0
  AST Above, Month 1 | 0 | 1 | 2 | 1
  AST Below, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  AST Below, Month 7 | 0 | 0 | 0 | 0
  AST Above, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  AST Above, Month 7 | 0 | 0 | 0 | 0
  HC Below, Month 1 | 0 | 6 | 2 | 4
  HC Above, Month 1 | 0 | 0 | 0 | 0
  HC Below, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  HC Below, Month 7 | 3 | 3 | 3 | 3
  HC Above, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  HC Above, Month 7 | 0 | 0 | 0 | 0
  NEU Below, Month 1 | 1 | 0 | 0 | 1
  NEU Above, Month 1 | 0 | 0 | 0 | 0
  NEU Below, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  NEU Below, Month 7 | 0 | 1 | 0 | 1
  NEU Above, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  NEU Above, Month 7 | 0 | 0 | 0 | 2
  Platelet Below, Month 1 | 0 | 0 | 0 | 0
  Platelet Above, Month 1 | 0 | 1 | 2 | 0
  Platelet Below, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  Platelet Below, Month 7 | 0 | 0 | 0 | 0
  Platelet Above, Month 7: number analyzed (Participants) | 16 | 18 | 18 | 20
  Platelet Above, Month 7 | 0 | 0 | 0 | 0

17. Secondary Outcome: Titers for DEN Neutralizing Antibodies Types 1, 2, 3 and 4
Description: as for outcome 3
Time Frame: At Month 0 and Month 1
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: ED50
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 18 | 19
ED50
  DEN-1, Month 0 | 10 [5 to 22] | 10 [4 to 24] | 13 [4 to 41] | 7 [4 to 12]
  DEN-1, Month 1 | 51 [15 to 179] | 20 [8 to 50] | 127 [36 to 450] | 7 [3 to 14]
  DEN-2, Month 0 | 9 [5 to 17] | 11 [4 to 26] | 11 [4 to 29] | 7 [4 to 10]
  DEN-2, Month 1 | 230 [84 to 630] | 94 [34 to 261] | 287 [95 to 870] | 7 [4 to 10]
  DEN-3, Month 0 | 8 [5 to 14] | 11 [5 to 25] | 10 [4 to 25] | 6 [4 to 9]
  DEN-3, Month 1 | 41 [13 to 124] | 22 [10 to 51] | 43 [14 to 135] | 6 [4 to 10]
  DEN-4, Month 0 | 9 [5 to 19] | 8 [4 to 16] | 10 [4 to 23] | 6 [4 to 7]
  DEN-4, Month 1 | 59 [16 to 224] | 52 [16 to 173] | 63 [17 to 238] | 6 [5 to 8]

18. Secondary Outcome: Number of Subjects With Antibody Titers Above the Assay Cut-off Value for Each DEN Serotype
Description: Assay cut-off values were greater than or equal to (≥) 10 estimated dose giving 50% (ED50) signal reduction when compared to a control without serum.
Time Frame: At Months 0, 1 and 7
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 18 | 19
Participants
  DEN-1, Month 0 | 4 | 3 | 3 | 1
  DEN-1, Month 1 | 11 | 9 | 13 | 1
  DEN-1, Month 7: number analyzed (Participants) | 16 | 18 | 15 | 19
  DEN-1, Month 7 | 15 | 14 | 13 | 2
  DEN-2, Month 0 | 4 | 3 | 3 | 3
  DEN-2, Month 1 | 18 | 15 | 16 | 2
  DEN-2, Month 7: number analyzed (Participants) | 16 | 18 | 15 | 19
  DEN-2, Month 7 | 16 | 15 | 15 | 2
  DEN-3, Month 0 | 4 | 4 | 3 | 1
  DEN-3, Month 1 | 12 | 12 | 12 | 1
  DEN-3, Month 7: number analyzed (Participants) | 16 | 18 | 15 | 19
  DEN-3, Month 7 | 12 | 13 | 13 | 2
  DEN-4, Month 0 | 4 | 3 | 3 | 1
  DEN-4, Month 1 | 10 | 12 | 11 | 3
  DEN-4, Month 7: number analyzed (Participants) | 16 | 18 | 15 | 19
  DEN-4, Month 7 | 13 | 14 | 11 | 1

19. Secondary Outcome: Number of Subjects With Antibody Titers Above the Assay Cut-off Value (Tetravalent Response) for All Dengue Serotypes
Description: The antibody titers and pre-vaccination status were determined by MN50 with a cut-off value equal to 1:10.
Time Frame: At Months 1 and 7
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 16 | 16 | 15 | 16
Participants
  Unprimed, Month 1: number analyzed (Participants) | 16 | 16 | 15 | 0
  Unprimed, Month 1 | 6 | 6 | 6 | 0
  Unprimed, Month 7: number analyzed (Participants) | 14 | 15 | 12 | 0
  Unprimed, Month 7 | 10 | 9 | 8 | 0
  Primed, Month 1: number analyzed (Participants) | 4 | 4 | 3 | 3
  Primed, Month 1 | 4 | 3 | 3 | 1
  Primed, Month 7: number analyzed (Participants) | 2 | 3 | 3 | 3
  Primed, Month 7 | 2 | 3 | 3 | 1

20. Secondary Outcome: Number of Subjects With Sero-response to Each DEN Type
Description: Sero-response defined as: For initially seronegative subjects (antibody titer < 10 ED50 for neutralizing antibodies to DEN 1, DEN 2, DEN 3, DEN 4 prior to vaccination), antibody titer ≥ 10 ED50 at post-vaccination; For initially seropositive subjects (antibody titer ≥ 10 ED50 for neutralizing antibodies to DEN 1, DEN 2, DEN 3, DEN 4 prior to vaccination), antibody titer at post-vaccination ≥ 4 fold the pre-vaccination antibody titer.
Time Frame: At Months 1 and 7
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
Number analyzed (Participants) | 20 | 20 | 18 | 19
Participants
  DEN-1, Month 1 | 10 | 6 | 10 | 0
  DEN-1, Month 7: number analyzed (Participants) | 16 | 18 | 15 | 19
  DEN-1, Month 7 | 14 | 11 | 10 | 1
  DEN-2, Month 1 | 16 | 13 | 14 | 0
  DEN-2, Month 7: number analyzed (Participants) | 16 | 18 | 15 | 19
  DEN-2, Month 7 | 14 | 13 | 13 | 0
  DEN-3, Month 1 | 11 | 8 | 10 | 0
  DEN-3, Month 7: number analyzed (Participants) | 16 | 18 | 15 | 19
  DEN-3, Month 7 | 11 | 11 | 11 | 1
  DEN-4, Month 1 | 9 | 10 | 9 | 2
  DEN-4, Month 7: number analyzed (Participants) | 16 | 18 | 15 | 19
  DEN-4, Month 7 | 12 | 12 | 9 | 0

21. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: as for outcome 1
Time Frame: During the 21-day (Days 0-20) follow-up after the study vaccine booster dose
Population: The analysis was performed on the Booster Total Vaccinated Cohort, which included all vaccinated subjects (with documented booster dose administration) with the symptom sheet filled in and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group
Number analyzed (Participants) | 8 | 12
Participants
  Any Pain | 0 | 0
  Grade 3 Pain | 0 | 0
  Any Redness | 1 | 2
  Grade 3 Redness | 0 | 0
  Any Swelling | 0 | 1
  Grade 3 Swelling | 0 | 0

22. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were abdominal pain, arthralgia, fatigue, fever [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)], headache, muscle aches, nausea, pain behind the eyes, photophobia, pruritus, rash and vomiting. Any = occurrence of the symptom regardless of intensity grade or relation to vaccination. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = oral fever > 39.0 °C. Related = symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 21-day (Days 0-20) follow-up after the study vaccine booster dose
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group
Number analyzed (Participants) | 8 | 12
Participants
  Any Abdominal pain | 0 | 1
  Grade 3 Abdominal pain | 0 | 0
  Related Abdominal pain | 0 | 0
  Any Arthralgia | 0 | 0
  Grade 3 Arthralgia | 0 | 0
  Related Arthralgia | 0 | 0
  Any Fatigue | 1 | 0
  Grade 3 Fatigue | 0 | 0
  Related Fatigue | 1 | 0
  Any Fever | 3 | 0
  Grade 3 Fever | 0 | 0
  Related Fever | 2 | 0
  Any Headache | 2 | 0
  Grade 3 Headache | 0 | 0
  Related Headache | 2 | 0
  Any Muscle aches | 0 | 0
  Grade 3 Muscle aches | 0 | 0
  Related Muscle aches | 0 | 0
  Any Nausea | 1 | 1
  Grade 3 Nausea | 0 | 0
  Related Nausea | 0 | 0
  Any Pain behind eyes | 0 | 0
  Grade 3 Pain behind eyes | 0 | 0
  Related Pain behind eyes | 0 | 0
  Any Photophobia | 0 | 1
  Grade 3 Photophobia | 0 | 0
  Related Photophobia | 0 | 1
  Any Pruritus | 0 | 0
  Grade 3 Pruritus | 0 | 0
  Related Pruritus | 0 | 0
  Any Rash | 0 | 0
  Grade 3 Rash | 0 | 0
  Related Rash | 0 | 0
  Any Vomiting | 1 | 0
  Grade 3 Vomiting | 0 | 0
  Related Vomiting | 0 | 0

23. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited AEs
Description: as for outcome 10
Time Frame: During the 31-day (Days 0-30) follow-up after the study vaccine booster dose
Population: The analysis was performed on the Booster Total Vaccinated Cohort, which included all vaccinated subjects (with documented booster dose administration) for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group
Number analyzed (Participants) | 9 | 12
Participants
  Any AE(s) | 6 | 3
  Grade 3 AE(s) | 2 | 0
  Related AE(s) | 0 | 1

24. Secondary Outcome: Number of Subjects With SAEs
Description: as for outcome 11
Time Frame: During the whole booster phase of the study (from pre-vaccination up to Month 6 post-vaccination with the booster dose)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group
Number analyzed (Participants) | 9 | 12
Participants | 2 | 0

25. Secondary Outcome: Number of Subjects With Hematological and Biochemical Determinations Within and Outside the Normal Ranges
Description: Among assessed haematological and biochemical parameters were: Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), hematocrit (HC), absolute neutrophil count (NEU) and platelet count (Platelet). Below = value below the laboratory reference range defined for the specified visit and laboratory parameter; Within = value within the laboratory reference range defined for the specified visit and laboratory parameter; Above = value above the laboratory reference range defined for the specified visit and laboratory parameter. Note: No blood sample was taken for these laboratory tests at Month 6 post-booster vaccination.
Time Frame: At each booster phase visit [pre-booster vaccination (PRE), study Visit 12 post-booster vaccination (Days 2, 5, 8 or 12) (FU1), study Visit 13 post-booster vaccination (Days 5, 8, 12 or 14) (FU2) and at Months 1 and 6 post-booster vaccination]
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group
Number analyzed (Participants) | 9 | 12
Participants
  ALT Within, PRE | 9 | 12
  ALT Within, FU1 | 9 | 12
  ALT Within, FU2 | 9 | 12
  ALT Within, Month 1 | 9 | 12
  ALT Below, PRE | 0 | 0
  ALT Below, FU1 | 0 | 0
  ALT Below, FU2 | 0 | 0
  ALT Below, Month 1 | 0 | 0
  ALT Above, PRE | 0 | 0
  ALT Above, FU1 | 0 | 0
  ALT Above, FU2 | 0 | 0
  ALT Above, Month 1 | 0 | 0
  AST Within, PRE | 9 | 12
  AST Within, FU1 | 9 | 12
  AST Within, FU2 | 9 | 12
  AST Within, Month 1 | 9 | 12
  AST Below, PRE | 0 | 0
  AST Below, FU1 | 0 | 0
  AST Below, FU2 | 0 | 0
  AST Below, Month 1 | 0 | 0
  AST Above, PRE | 0 | 0
  AST Above, FU1 | 0 | 0
  AST Above, FU2 | 0 | 0
  AST Above, Month 1 | 0 | 0
  HC Within, PRE | 8 | 10
  HC Within, FU1 | 8 | 9
  HC Within, FU2 | 8 | 11
  HC Within, Month 1 | 8 | 12
  HC Below, PRE | 1 | 2
  HC Below, FU1 | 1 | 3
  HC Below, FU2 | 1 | 1
  HC Below, Month 1 | 1 | 0
  HC Above, PRE | 0 | 0
  HC Above, FU1 | 0 | 0
  HC Above, FU2 | 0 | 0
  HC Above, Month 1 | 0 | 0
  NEU Within, PRE | 9 | 11
  NEU Within, FU1 | 8 | 12
  NEU Within, FU2 | 8 | 12
  NEU Within, Month 1 | 7 | 12
  NEU Below, PRE | 0 | 0
  NEU Below, FU1 | 1 | 0
  NEU Below, FU2 | 0 | 0
  NEU Below, Month 1 | 2 | 0
  NEU Above, PRE | 0 | 1
  NEU Above, FU1 | 0 | 0
  NEU Above, FU2 | 1 | 0
  NEU Above, Month 1 | 0 | 0
  Platelet Within, PRE | 9 | 12
  Platelet Within, FU1 | 9 | 12
  Platelet Within, FU2 | 9 | 12
  Platelet Within, Month 1 | 8 | 12
  Platelet Below, PRE | 0 | 0
  Platelet Below, FU1 | 0 | 0
  Platelet Below, FU2 | 0 | 0
  Platelet Below, Month 1 | 0 | 0
  Platelet Above, PRE | 0 | 0
  Platelet Above, FU1 | 0 | 0
  Platelet Above, FU2 | 0 | 0
  Platelet Above, Month 1 | 1 | 0

26. Secondary Outcome: Number of Subjects With Alert Values for Safety Laboratory Determinations
Description: as for outcome 12
Time Frame: During the 31-day (Days 0-30) follow-up after the study vaccine booster dose
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group
Number analyzed (Participants) | 9 | 12
Participants
  ALT | 0 | 0
  AST | 0 | 0
  HC | 0 | 0
  NEU | 0 | 0
  Platelet | 0 | 0

27. Secondary Outcome: Number of Subjects With Abnormal Findings at Dengue Physical Examination
Description: The abnormal findings at Dengue physical examination included: Conjunctival hemorrhage, Conjunctival injection, Generalized lymphadenopathy, Generalized rash, Hepatomegaly, Lymphadenopathy, Mucosal hemorrhage, Rash, Skin hemorrhage and Splenomegaly. Rash involved < 50% of the body surface; Generalized rash involved at least 50% of the body surface. Generalized lymphadenopathy was defined as palpable lymph nodes in four or more of the following locations: cervical, axillary, inguinal or other, with right and left sides considered as separate locations. Note: Results only available during the 31-day follow-up period (Month 1) after the booster dose, instead of at each booster phase visit [pre-vaccination, study Visit 12 post-booster vaccination (Days 2, 5, 8 or 12), Visit 13 post-booster vaccination (Days 5, 8, 12 or 14) and at Months 1 and 6 post-booster vaccination].
Time Frame: At Month 1 post-booster vaccination
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group
Number analyzed (Participants) | 9 | 12
Participants
  Conjunctival hemorrhage | 0 | 0
  Conjunctival injection | 0 | 0
  Generalized lymphadenopathy | 0 | 0
  Generalized rash | 0 | 0
  Hepatomegaly | 0 | 2
  Lymphadenopathy | 1 | 2
  Mucosal hemorrhage | 1 | 0
  Rash | 0 | 0
  Skin hemorrhage | 0 | 0
  Splenomegaly | 0 | 0

28. Secondary Outcome: Number of Subjects With Suspected and Confirmed Dengue
Description: The number of subjects with suspected and confirmed Dengue post-booster vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up after the study vaccine booster dose
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group
Number analyzed (Participants) | 9 | 12
Participants
  Suspected dengue | 0 | 0
  Confirmed dengue | 0 | 0

29. Secondary Outcome: Number of Subjects With Measurable Dengue Viremia
Description: The number of subjects with measurable dengue viremia at specified timepoints.
Time Frame: At study Visit 12 (Days 2, 5, 8 or 12) (FU1), study Visit 13 post-booster vaccination (Days 5, 8, 12 or 14) (FU2) and at study Visit 14 (Month 1 post-booster vaccination)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group
Number analyzed (Participants) | 9 | 12
Participants
  DEN-1 Positive, FU1 | 0 | 0
  DEN-2 Positive, FU1 | 0 | 0
  DEN-3 Positive, FU1 | 0 | 0
  DEN-4 Positive, FU1 | 0 | 0
  DEN-1 Positive, FU2 | 0 | 0
  DEN-2 Positive, FU2 | 0 | 0
  DEN-3 Positive, FU2 | 0 | 0
  DEN-4 Positive, FU2 | 0 | 0
  DEN-1 Positive, Month 1 | 0 | 0
  DEN-2 Positive, Month 1 | 0 | 1
  DEN-3 Positive, Month 1 | 0 | 0
  DEN-4 Positive, Month 1 | 0 | 0

30. Secondary Outcome: Number of Subjects With Antibody Titers Above the Assay Cut-off Value for Each DEN Serotype
Description: Assay cut-off values were greater than or equal to (≥) 10 estimated dose giving 50% (ED50) signal reduction when compared to a control without serum. Not primed = Not primed by MN50; Primed = Primed by MN50. Primed subject is a subject with neutralizing antibody titer ≥ 10 ED50 at pre-vaccination for at least one DEN type. Not primed subject is a subject with neutralizing antibody titer <10 ED50 for any DEN type at pre-vaccination.
Time Frame: Before (PRE) and one month after the booster vaccination (Month 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group
Number analyzed (Participants) | 6 | 7
Participants
  DEN-1 Not primed, PRE | 4 | 5
  DEN-1 Not primed, Month 1 | 5 | 7
  DEN-1 Primed, PRE: number analyzed (Participants) | 2 | 2
  DEN-1 Primed, PRE | 2 | 2
  DEN-1 Primed, Month 1: number analyzed (Participants) | 2 | 2
  DEN-1 Primed, Month 1 | 2 | 2
  DEN-2 Not primed, PRE | 4 | 4
  DEN-2 Not primed, Month 1 | 5 | 7
  DEN-2 Primed, PRE: number analyzed (Participants) | 2 | 2
  DEN-2 Primed, PRE | 2 | 2
  DEN-2 Primed, Month 1: number analyzed (Participants) | 2 | 2
  DEN-2 Primed, Month 1 | 2 | 2
  DEN-3 Not primed, PRE | 1 | 3
  DEN-3 Not primed, Month 1 | 5 | 4
  DEN-3 Primed, PRE: number analyzed (Participants) | 2 | 2
  DEN-3 Primed, PRE | 2 | 2
  DEN-3 Primed, Month 1: number analyzed (Participants) | 2 | 2
  DEN-3 Primed, Month 1 | 2 | 2
  DEN-4 Not primed, PRE | 2 | 3
  DEN-4 Not primed, Month 1 | 5 | 4
  DEN-4 Primed, PRE: number analyzed (Participants) | 2 | 2
  DEN-4 Primed, PRE | 2 | 2
  DEN-4 Primed, Month 1: number analyzed (Participants) | 2 | 2
  DEN-4 Primed, Month 1 | 2 | 2

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 21-day (Days 0-20) follow up period after primary vaccination; Unsolicited AEs: during the 31-day (Days 0-30) follow up period after primary vaccination; SAEs: throughout the whole study period (from Day 0 up to Month 6 post-booster vaccination).
Arm/Group | Dengue Formulation 17a Group | Dengue Formulation 17b Group | Dengue Formulation 19 Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 1/22 | 1/21 | 1/21
Other Adverse Events (participants affected / at risk) | 20/22 | 19/22 | 18/21 | 16/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Dengue Formulation 17a Group (N=22) | Dengue Formulation 17b Group (N=22) | Dengue Formulation 19 Group (N=21) | Placebo Group (N=21)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Primary phase
Physical assault (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Primary phase
Procedural hypertention (Injury, poisoning and procedural complications) | 0 (0) | 1/9 | 0/12 (0) | 0 (0) — Booster phase
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1/9 | 0/12 (0) | 0 (0) — Booster phase
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dengue Formulation 17a Group (N=22) | Dengue Formulation 17b Group (N=22) | Dengue Formulation 19 Group (N=21) | Placebo Group (N=21)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 5 (6) | 4 (4) | 4 (5)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4) | 3 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 8 (9) | 3 (3) | 5 (6) | 6 (7)
Eye pain (Eye disorders) | 4 (5) | 7 (8) | 5 (6) | 3 (3)
Fatigue (General disorders) | 10 (12) | 8 (10) | 6 (8) | 7 (10)
Headache (Nervous system disorders) | 14 (19) | 9 (13) | 10 (11) | 9 (14)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (6) | 4 (4) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 4 (6) | 3 (3) | 2 (2)
Pain (General disorders) | 9 (14) | 3 (3) | 5 (5) | 5 (7)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 4 (4) | 3 (3) | 4 (4) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (10) | 3 (3) | 3 (3) | 4 (6)
Pyrexia (General disorders) | 5 (5) | 4 (4) | 3 (3) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 3 (3) | 3 (3) | 0 (0)
Swelling (General disorders) | 7 (7) | 5 (5) | 5 (5) | 3 (3)
Vessel puncture site haemorrhage (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.